CLINICAL TRIAL: NCT00743548
Title: Comparison of Inter-dental Brush to Dental Floss for Reduction of Plaque and Bleeding in Areas With Intact Papilla: A Clinical Trial
Brief Title: Comparing the Inter-dental Brush to Dental Floss
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Foundation for Dental Hygiene Research and Education (Other); British Columbia Dental Hygienists' Association (BCDHA) (Industry); Curaden Swiss (Industry)
Responsible Party: Pauline Imai, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: H08-01078
Record Dates: First submitted 2008-08-27; First posted 2008-08-29 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Gingivitis
Keywords: interdental self-care aids; plaque; bleeding gums
MeSH Terms: conditions — Gingivitis; Plaque, Amyloid; Gingival Hemorrhage

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Interdental brush (IB), the intervention is a small multi-tufted brush on a wire attached to a long angled handle that is inserted in a horizontal plane between the teeth. The IB is inserted once and removed.
  Interventions: Device: IB = Interdental brush, the intervention
- 2 (Placebo Comparator): Dental floss (DF), the positive control, is waxed dental floss; nylon covered with a water soluble unflavoured wax to facilitate easier access the contact points of teeth. DF is rubbed against the interproximal surfaces of the teeth 2-4 times on each surface.
  Interventions: Device: DF = Dental floss, the positive control

INTERVENTIONS:
Device: IB = Interdental brush, the intervention — IB is a small multi-tufted brush on a wire attached to a long angled handle that is inserted in a horizontal plane between the teeth. The IB is inserted once and removed.
  Arms: 1
Device: DF = Dental floss, the positive control — DF is waxed dental floss; nylon covered with a water soluble unflavoured wax to facilitate easier access the contact points of teeth. DF is rubbed against the interproximal surfaces of the teeth 2-4 times on each surface.
  Arms: 2

SUMMARY:
The study's purpose is to find an easy and effective alternative to dental floss for those persons who cannot or choose not to dental floss so that they can maintain and/or achieve optimal oral health. The study hypothesis is that the inter-dental brush is as effective as dental floss for removing plaque from between the teeth and for reducing bleeding gums in persons with gingivitis, but may be easier to use and thus encourage daily home use.

DETAILED DESCRIPTION:
Purpose:

To determine if the interdental brush is just as effective at removing plaque and reducing bleeding gums between the teeth as dental floss.

Rationale:

Many people find dental floss difficult to use and thus, do not floss daily to maintain oral health and prevent gum disease. These individuals may find the interdental brush easier to use and may be motivated to use it daily for optimal oral health.

Study design:

Study subjects will use the dental floss AND the interdental brush for 12 weeks. Plaque and bleeding scores will be measured before the study begins (week 0), mid-way (week 6), and at the end of the 12 weeks. All study subjects receive a teeth cleaning prior to the first measurements and oral hygiene instructions on how to floss and use the interdental brush. Subjects will also answer 4 short questions about their product preference and ease of use.

Study subjects:

32 healthy adult volunteers with bleeding gums. To be included in the study, subjects require 8 bleeding sites, 4 areas that can accommodate the interdental brush, dexterity to dental floss, and willingness to come for 4 study visits. Exclusion criteria include smokers because this can affect the bleeding scores; individuals with braces (orthodontia) which affects plaque levels; individuals using chlorhexidine which is a prescription strength mouthwash used to treat moderate to severe gum disease; pregnant women; and those individuals requiring antibiotics prior to dental appointments. Enrolled study subjects receive a teeth cleaning (value $180), $75 for completing the study, and all study related supplies.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Minimum of 4 interproximal areas that can accommodate a minimum 0.6 mm interdental brush width
* Minimum of 8 interproximal bleeding sites upon stimulation
* Dexterity to use manual waxed dental floss
* Able to attend all 4 study visits

Exclusion Criteria:

* Require premedication with antibiotics prior to dental therapy
* Use chlorhexidine or over-the-counter mouthwash during the study
* Smoke
* Have orthodontia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Plaque and bleeding reduction | 12 weeks

SECONDARY OUTCOMES:
Product preference between dental floss and interdental brush | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Imai, MSc., Principal Investigator — University of British Columbia; Penny Hatzimanolakis, Study Director — University of British Columbia
Locations (1):
- University of British Columbia Nobel Biocare Oral Health Centre, Vancouver, British Columbia, Canada